CLINICAL TRIAL: NCT06010485
Title: The Effect of Serial Casting and Physical Therapy on Ankle Range of Motion, Toe Walking Severity, Walking Balance, Functional Health Related Quality of Life in Children With Idiopathic Toe Walking
Brief Title: The Effect of Serial Casting and Physical Therapy in Children With Idiopathic Toe Walking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: illeezozge
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Idiopathic Toe Walking
Keywords: Idiopathic Toe Walking; Serial Casting; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, single blinded, controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Serial Casting (Active Comparator): The serial casting group received intermittent serial casting once every three days for three weeks.
  Interventions: Other: Serial Casting
- Exercise (Active Comparator): The physical therapy group underwent three sessions per week for three weeks, consisting of stretching exercises, strengthening exercises, balance training, proprioception exercises, and walking on heels.
  Interventions: Other: Exercise
- Control Group (No Intervention): This group consists of the patients on the waitlist.

INTERVENTIONS:
Other: Serial Casting — A short leg cast is applied to the serial casting group by an orthopedic specialist once every three days for three weeks.
  Arms: Serial Casting
Other: Exercise — Stretching exercises, strengthening exercises, balance exercises, proprioception exercises, and heel walking exercises are applied to the physical therapy group for 3 weeks with a physiotherapist for 3 sessions a week.
  Arms: Exercise

SUMMARY:
Children who continue to walk on their tiptoes after developing a heel-toe gait normally are diagnosed with idiopathic toe walking (ITW). The study's aim was to investigate the effects of serial casting and physical therapy on joint range of motion (ROM), toe walking severity, functional health and health-related quality of life, walking balance, and satisfaction from treatment in ITW, in comparison with the control group.

DETAILED DESCRIPTION:
Children with ITW aged 3-10 years are randomized into three groups: the serial casting group (n=10), the physical therapy group (n=10), and the wait-list control group (n=10). Patients with ankle contracture and previous interventions are excluded. The serial casting group is planned to receive intermittent serial casting once every three days for three weeks. The physical therapy group is planned to undergo three sessions per week for three weeks, consisting of stretching exercises, strengthening exercises, balance training, proprioception exercises, and walking on heels. The patients were assessed by blinded investigators at before treatment (BT), post-treatment (PT: 3th week), 1st month (1MPT), 3rd months (3MPT), and 6th months post-treatment (6MPT). To ensure ethical considerations, only control group was followed-up until the 1MPT.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 3-10 years
2. Patients with idiopathic toe walking diagnosis
3. To be evaluated by a pediatric neurologist, not to have abnormal findings in cranial and all spinal magnetic resonance imaging and electrophysiological examinations performed when deemed necessary, and creatinine kinase values are within normal limits ((Absence of any neurological, orthopedic or psychiatric pathology to explain the toe walking pattern (cerebral palsy, neuropathy, myopathy, autism, developmental disorders, etc.)

Exclusion Criteria:

1. Have previously conservative or surgical treatment
2. Presence of plantar flexion contracture

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Range of Motion (ROM) | Day 0
  Ankle dorsiflexion ROM with extended knee
Range of Motion (ROM) | 3rd week
  Ankle dorsiflexion ROM with extended knee
Range of Motion (ROM) | 7th week
  Ankle dorsiflexion ROM with extended knee
Range of Motion (ROM) | 15th week
  Ankle dorsiflexion ROM with extended knee
Range of Motion (ROM) | 27th week
  Ankle dorsiflexion ROM with extended knee
Range of Motion (ROM) | Day 0
  Ankle dorsiflexion ROM with flexed knee
Range of Motion (ROM) | 3rd week
  Ankle dorsiflexion ROM with flexed knee
Range of Motion (ROM) | 7th week
  Ankle dorsiflexion ROM with flexed knee
Range of Motion (ROM) | 15th week
  Ankle dorsiflexion ROM with flexed knee
Range of Motion (ROM) | 27th week
  Ankle dorsiflexion ROM with flexed knee
Toe Walking Severity Scale | Day 0
  The family is asked how long the child tiptoe walks during the day. The evaluation is as follows.
  Stage 1: Toe walking 76-100% of the time Stage 2: Toe walking 51-75% of the time Stage 3: Toe walking 26-50% of the time Stage 4: Toe walking 10-25% of the time Stage 5: Sole pressing but early heel lift (occasional toe gait <10%) Stage 6: Normal heel strike
Toe Walking Severity Scale | 3rd week
  The family is asked how long the child tiptoe walks during the day. The evaluation is as follows.
  Stage 1: Toe walking 76-100% of the time Stage 2: Toe walking 51-75% of the time Stage 3: Toe walking 26-50% of the time Stage 4: Toe walking 10-25% of the time Stage 5: Sole pressing but early heel lift (occasional toe gait <10%) Stage 6: Normal heel strike
Toe Walking Severity Scale | 7th week
  The family is asked how long the child tiptoe walks during the day. The evaluation is as follows.
  Stage 1: Toe walking 76-100% of the time Stage 2: Toe walking 51-75% of the time Stage 3: Toe walking 26-50% of the time Stage 4: Toe walking 10-25% of the time Stage 5: Sole pressing but early heel lift (occasional toe gait <10%) Stage 6: Normal heel strike
Toe Walking Severity Scale | 15th week
  The family is asked how long the child tiptoe walks during the day. The evaluation is as follows.
  Stage 1: Toe walking 76-100% of the time Stage 2: Toe walking 51-75% of the time Stage 3: Toe walking 26-50% of the time Stage 4: Toe walking 10-25% of the time Stage 5: Sole pressing but early heel lift (occasional toe gait <10%) Stage 6: Normal heel strike
Toe Walking Severity Scale | 27th week
  The family is asked how long the child tiptoe walks during the day. The evaluation is as follows.
  Stage 1: Toe walking 76-100% of the time Stage 2: Toe walking 51-75% of the time Stage 3: Toe walking 26-50% of the time Stage 4: Toe walking 10-25% of the time Stage 5: Sole pressing but early heel lift (occasional toe gait <10%) Stage 6: Normal heel strike

SECONDARY OUTCOMES:
Pediatric Outcomes Data Collection Instrument (PODCI) | Day 0
  PODCI evaluates functional health status through an 86 item questionnaire. Scoring varies greatly due to the multiple weighted scores of some items, scores range from 0-3 for some items and 0-6 for others. The overall score comes from 4 functional assessment scores, a global function score, and a happiness score. These scores range from 0-100 with lower scores representing higher levels of disability.
Pediatric Outcomes Data Collection Instrument (PODCI) | 3rd week
  PODCI evaluates functional health status through an 86 item questionnaire. Scoring varies greatly due to the multiple weighted scores of some items, scores range from 0-3 for some items and 0-6 for others. The overall score comes from 4 functional assessment scores, a global function score, and a happiness score. These scores range from 0-100 with lower scores representing higher levels of disability.
Pediatric Outcomes Data Collection Instrument (PODCI) | 7th week
  PODCI evaluates functional health status through an 86 item questionnaire. Scoring varies greatly due to the multiple weighted scores of some items, scores range from 0-3 for some items and 0-6 for others. The overall score comes from 4 functional assessment scores, a global function score, and a happiness score. These scores range from 0-100 with lower scores representing higher levels of disability.
Pediatric Outcomes Data Collection Instrument (PODCI) | 15th week
  PODCI evaluates functional health status through an 86 item questionnaire. Scoring varies greatly due to the multiple weighted scores of some items, scores range from 0-3 for some items and 0-6 for others. The overall score comes from 4 functional assessment scores, a global function score, and a happiness score. These scores range from 0-100 with lower scores representing higher levels of disability.
Pediatric Outcomes Data Collection Instrument (PODCI) | 27th week
  PODCI evaluates functional health status through an 86 item questionnaire. Scoring varies greatly due to the multiple weighted scores of some items, scores range from 0-3 for some items and 0-6 for others. The overall score comes from 4 functional assessment scores, a global function score, and a happiness score. These scores range from 0-100 with lower scores representing higher levels of disability.
Tandem Walk Test | Day 0
  The participants are asked to walk in a straight line with one foot just in front of the other (heel to toe), arms at their sides.
Tandem Walk Test | 3rd week
  The participants are asked to walk in a straight line with one foot just in front of the other (heel to toe), arms at their sides.
Tandem Walk Test | 7th week
  The participants are asked to walk in a straight line with one foot just in front of the other (heel to toe), arms at their sides.
Tandem Walk Test | 15th week
  The participants are asked to walk in a straight line with one foot just in front of the other (heel to toe), arms at their sides.
Tandem Walk Test | 27th week
  The participants are asked to walk in a straight line with one foot just in front of the other (heel to toe), arms at their sides.
Visual Analog Scale | 3rd week
  All participants are asked about satisfaction with treatment through a smiley face visual analog scale 'smiley face' visual analogue scale (0-10, 0 for full satisfaction)
Visual Analog Scale | 7th week
  All participants are asked about satisfaction with treatment through a smiley face visual analog scale 'smiley face' visual analogue scale (0-10, 0 for full satisfaction)
Visual Analog Scale | 15th week
  All participants are asked about satisfaction with treatment through a smiley face visual analog scale 'smiley face' visual analogue scale (0-10, 0 for full satisfaction)
Visual Analog Scale | 27th week
  All participants are asked about satisfaction with treatment through a smiley face visual analog scale 'smiley face' visual analogue scale (0-10, 0 for full satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Esra Giray, Principal Investigator — Fatih Sultan Mehmet training and Research Hospital, Istanbul-Turkey
Locations (1):
- Fatih Sultan Mehmet Trainig and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pomarino D, Ramirez Llamas J, Martin S, Pomarino A. Literature Review of Idiopathic Toe Walking: Etiology, Prevalence, Classification, and Treatment. Foot Ankle Spec. 2017 Aug;10(4):337-342. doi: 10.1177/1938640016687370. Epub 2017 Jan 16. PMID 28092971
- [Background] Engelbert R, Gorter JW, Uiterwaal C, van de Putte E, Helders P. Idiopathic toe-walking in children, adolescents and young adults: a matter of local or generalised stiffness? BMC Musculoskelet Disord. 2011 Mar 21;12:61. doi: 10.1186/1471-2474-12-61. PMID 21418634
- [Background] Herrin K, Geil M. A comparison of orthoses in the treatment of idiopathic toe walking: A randomized controlled trial. Prosthet Orthot Int. 2016 Apr;40(2):262-9. doi: 10.1177/0309364614564023. Epub 2015 Jan 27. PMID 25628380
- [Background] Pomarino D, Ramirez Llamas J, Pomarino A. Idiopathic Toe Walking: Family Predisposition and Gender Distribution. Foot Ankle Spec. 2016 Oct;9(5):417-22. doi: 10.1177/1938640016656780. Epub 2016 Jul 1. PMID 27370652
- [Background] Satila H, Beilmann A, Olsen P, Helander H, Eskelinen M, Huhtala H. Does Botulinum Toxin A Treatment Enhance the Walking Pattern in Idiopathic Toe-Walking? Neuropediatrics. 2016 Jun;47(3):162-8. doi: 10.1055/s-0036-1582138. Epub 2016 Apr 18. PMID 27089542
- [Background] Engstrom P, Bartonek A, Tedroff K, Orefelt C, Haglund-Akerlind Y, Gutierrez-Farewik EM. Botulinum toxin A does not improve the results of cast treatment for idiopathic toe-walking: a randomized controlled trial. J Bone Joint Surg Am. 2013 Mar 6;95(5):400-7. doi: 10.2106/JBJS.L.00889. PMID 23467862
- [Background] Williams CM, Tinley P, Curtin M. The Toe Walking Tool: a novel method for assessing idiopathic toe walking children. Gait Posture. 2010 Oct;32(4):508-11. doi: 10.1016/j.gaitpost.2010.07.011. Epub 2010 Aug 7. PMID 20692159
- [Derived] Giray E, Akpinar P, Illeez OG, Kahraman HC, Kocibar M, Kutsal A, Hacifazlioglu NE, Uyur E, Unlu Ozkan F, Aktas I, Yilmaz B, Karadag-Saygi E. A comparative randomized-controlled trial of serial casting and exercises on ankle range of motion, toe walking severity, walking balance, and functional health-related quality of life in children with idiopathic toe walking. J Pediatr Orthop B. 2025 Sep 1;34(5):465-476. doi: 10.1097/BPB.0000000000001250. Epub 2025 Jul 29. PMID 40167594